CLINICAL TRIAL: NCT04313465
Title: Troponin-only Manchester Acute Coronary Syndromes Decision Aid to Reduce Unnecessary Hospitalisation for Patients With Chest Pain: a Randomized, Controlled Point of Care Trial
Brief Title: T-MACS Decision Aid: a Randomized, Controlled Point of Care Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: CI no longer wishes to complete this study due to Covid-19
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R04799; 245543 (Other: IRAS Project ID)
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Heart Attack; Chest Pain; Acute Coronary Syndrome
Keywords: T-MACS
MeSH Terms: conditions — Myocardial Infarction; Chest Pain; Acute Coronary Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Routine Care) (No Intervention): Participants will undergo risk stratification using the T-MACS decision aid, which includes a cardiac troponin blood test upon admission to the Emergency Department. Participants will then have a repeat cardiac troponin blood test in 3 hours.
- Intervention (Immediate Discharge) (Experimental): Participants will undergo risk stratification using the T-MACS decision aid, which includes a troponin blood test upon admission to the Emergency Department. Participants will then be discharged.
  Interventions: Other: Immediate discharge

INTERVENTIONS:
Other: Immediate discharge — Participants discharged after initial blood test for cardiac troponin and risk stratification using the T-MACS decision aid
  Arms: Intervention (Immediate Discharge)

SUMMARY:
The aim of the study is to establish whether the safety of the T-MACS decision aid to immediately 'rule out' acute coronary syndromes with one blood sample for the cardiac damage marker troponin, is non-inferior to an approach requiring serial troponin sampling over three hours.

DETAILED DESCRIPTION:
We will conduct a randomized, controlled point of care trial embedded in routine practice. We will ask clinicians to obtain written informed consent during the course of their clinical duties. Patients who have suspected cardiac chest pain, who are identified as being at very low risk by the T-MACS algorithm, will be invited to participate.

Patients will then be randomly allocated to be advised that they can be discharged immediately (so long as the doctor and patient have no other concerns; this is the originally intended use of T-MACS; intervention arm) or to receive a second blood test after 3 hours (current practice; control arm).

Participants will then be followed up by electronic record review after 30 days and 12 months. Other than the difference in the requirement for a second blood test, participants will not notice any change to their care.

The accelerated pathway (involving a single blood test) has been shown to be safe in observational research involving over 5,000 patients. All of the data that are collected are the same of those that are collected in routine care, and they will be anonymised for analysis.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Presents to the Emergency Department with pain, discomfort or pressure in the chest, epigastrium, neck, jaw, or upper limb without an apparent non-cardiac source which the treating physician believes warrants investigation for possible acute coronary syndrome
* The patient is identified as being at 'very low risk' by the T-MACS decision aid following a single hs-cTn test at the time of arrival in the Emergency Department

Exclusion Criteria:

* No capacity to provide informed consent
* Inability to communicate in English language if translation services are unavailable
* Patient is a prisoner
* No NHS number (precluding electronic follow up)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
The incidence of major adverse cardiac event | 30 days
  This is defined as cardiovascular death or acute myocardial infarction (including prevalent acute myocardial infarction at the time of initial attendance)

SECONDARY OUTCOMES:
The incidence of coronary revascularization | 30 days
  If the participant has had a cardiac bypass or has had stents inserted to improve blood flow
Length of initial hospital stay | 30 days
  How long the participant was in hospital for after Emergency Department admission
The incidence of cardiovascular death or acute myocardial infarction | 1 year
  If the patient has had another cardiac episode, or if the participant has died due to a heart attack

CONTACTS AND LOCATIONS:
Overall Officials: Richard Body, Principal Investigator — Manchester University NHS Foundation Trust
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No